CLINICAL TRIAL: NCT01663246
Title: Cross-Sectional Study of Oral Health in Patients After Parotid-Sparing Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Avraham Eisbruch, Newman Family Professor of Radiation Oncology and Professor of Radiation, University of Michigan Rogel Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005.097; HUM00000970 (Other: University of Michigan Medical School IRB)
Record Dates: First submitted 2012-07-24; First posted 2012-08-13 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Adults (Active Comparator): Healthy adults over the age of 18, with no history of surgery to the salivary glands, or cancer therapy.
  Interventions: Procedure: Saliva Sample
- Radiation for Head and Neck Cancer (Active Comparator): History of radiation therapy for head and neck cancer.
  Interventions: Procedure: Saliva Sample

INTERVENTIONS:
Procedure: Saliva Sample — Small plastic cups will be placed on the inside of subject cheeks, and held in place with gentle suction. These cups are attached to tubes which will allow the collection of saliva into a test tube. Saliva will also be collected from the glands underneath the tongue using a small gentle suction device, similar to the one used by a dentist. Saliva production will be stimulated by dabbing a mild citric acid solution that tastes like lemon onto the tongue using a Q-Tip. After this test, subjects will also be asked to chew wax to simulate saliva, and the saliva that accumulates in their mouth will be collected by spitting into a test tube.

SUMMARY:
The investigators are conducting research about oral health and saliva to find out more about the impact of radiation therapy on the oral health of patients.

In order to better understand the role of saliva in maintaining oral health in these patients, the investigators will be collecting, storing, and analyzing the quality of saliva, including the protein content, collected from patients following radiation therapy as well as saliva collected from normal healthy adults.

DETAILED DESCRIPTION:
Radiation-induced xerostomia is the most common long term complication of head and neck radiation, is usually permanent and is the most frequent reason for reduced quality of life in these patients. The loss of antimicrobial, buffering, cleansing and remineralizing effects of saliva markedly increases the risk for dental caries. Extractions of diseased teeth located in irradiated bone and dental infection involving the bone can trigger osteoradionecrosis (ORN), another serious complication of high dose radiation of the jaws. Therefore, current dental treatment guidelines recommend the extraction of diseased teeth and any teeth that might require extraction in the future, before radiation therapy. (NCI, 1990; Rankin et al, 2003; NIDCR, 2005) As a result, patients with head and neck cancer often have many or all teeth extracted, especially those patients who are judged unlikely to comply with lifelong, daily topical fluoride, oral hygiene practices and frequent professional dental care. (Bruins et al, 1999)

ELIGIBILITY:
Inclusion Criteria:

* All subjects who have been enrolled in a parotid-sparing IMRT protocol for head and neck cancer at University of Michigan.
* At least 6 months has elapsed since the completion of RT, at the time of assessment for this study.
* All subjects must sign a University of Michigan Health System- IRB approved informed consent.
* Documented Karnofsky performance status > 60
* These subjects will all have American Joint Committee on Cancer (AJCC) Stage III or Stage IV disease. (Green et al, 2001) (Appendix 2); non-metastatic, curable disease

Exclusion Criteria:

* History of surgical removal of major salivary gland(s).
* Patients edentulous prior to radiation therapy.
* Pregnancy or lactation
* Patients residing in prison.
* Age< 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
prevalence of dental caries in patients after PS-IMRT | 24 Months
  Various surveys and questionnaires administered for data collection as well as potential risk indicators for dental caries. Oral examination and saliva specimins collected will determine acid, plaque and exposure to tobacco products
prevalence of tooth loss in patients after PS-IMRT | 24 months
  Various surveys and questionnaires administered for data collection as well as potential risk indicators for dental caries. Oral examination and saliva specimins collected will determine acid, plaque and exposure to tobacco products

SECONDARY OUTCOMES:
prevalence of periodontal disease after PS-IMRT | 24 Months
  number of caries in individual subjects will depend on number of teeth and/or surfaces at risk, we will need to report "prevalence" after adjusting for the total surfaces at risk for each patient. In addition, because data in the cross-sectional cohort will be obtained from patients at different follow-up times since RT, the relationship between prevalence and time since RT will need to be explored to take into account the time effect.

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Eisbruch, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States